CLINICAL TRIAL: NCT06147336
Title: A Multi-center, National, Open Label, Prospective Study to Evaluate the Safety, Usability and Performance of the V-LAP™ System, for Wirelessly Measuring and Monitoring Left Atrial Pressure (Lap) in Patients With Advanced CHF
Brief Title: A Multi-center, National, Open-label, Prospective Study to Evaluate the Performance of the V-Lap™ System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vectorious Medical Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLC-0035
Record Dates: First submitted 2023-11-19; First posted 2023-11-27 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- V-LAP™ System (Experimental): Heart failure subjects - Percutaneous implantation of the V-LAP™ implant by right heart catheterization (RHC) approach and daily LAP measurements at home and will be trained on the use of the device for self-management.
  Interventions: Device: V-LAP™ SYSTEM

INTERVENTIONS:
Device: V-LAP™ SYSTEM — Delivery of the V-LAP™ implant by right heart catheterization. A catheter-based approach in a trans-septal puncture procedure, fixated within the inter-atrial septum.

SUMMARY:
The objective of this study is to evaluate the safety and performance of the V-LAP System in subjects with New York Heart Association (NYHA) functional class II and III HF, irrespective of left ventricular ejection fraction.

DETAILED DESCRIPTION:
The V- LAP™ System is intended for wirelessly measuring and monitoring LAP. The V-LAP™ System is indicated for subjects with chronic symptomatic ACC/AHA Stage C subjects Heart Failure.

Pressure-guided medical management of study participants, with the goal of reducing hospitalizations and improving quality of life, will be implemented using a physician-directed patient self-management approach.

V-LAP-PSM (Patient Self-management), Patient Guidance Application is a smartphone application that guides the patient on how to self-adjust the treatment, according to physician prescription, and when to approach their healthcare provider (HCP).

Freedom from study (Device and/or system) related Major Adverse Cardiac and Neurological Events (MACNE as defined in the protocol) up to six months post-procedure, as adjudicated by the independent Clinical Events Committee.

ELIGIBILITY:
1. Ischemic or non-ischemic cardiomyopathy and documented heart failure for at least 6 months (diagnosis of HF ≥ 6 months), regardless of ejection fraction.
2. NYHA Class II heart failure (HF) subjects, documented at Baseline Visit regardless of ejection fraction, meeting both inclusion criteria in subsections (2a) and (2b) or NYHA Class III heart failure (HF) subjects, documented at Baseline Visit regardless of ejection fraction, meeting at least one inclusion criteria in subsections (2a) and (2b).

   1. Have a minimum of one (1) HF hospitalization or equivalent (HF Emergency Department Visit or HF Urgent Clinic Visit) within the last 12 months associated with signs/symptoms of congestion requiring treatment with intravenous (IV) diuretic. If Cardiac Resynchronization Therapy (CRT) device previously implanted, the HF hospitalization or equivalent must be ≥ 30 days after CRT implantation.
   2. Have a corrected* elevated outpatient Brain Natriuretic Peptide (BNP) level of at least 300 pg/ml or an N-terminal pro-BNP (NT-proBNP) level of at least 1,500 pg/ml, according to local measurement, within 90-days of the Baseline Visit.

      * Thresholds for NT-proBNP will be corrected for body mass index (BMI) using a 4% reduction per BMI unit over 20 kg/m2. If the subject is on ARNI, NT-proBNP should be used exclusively.
3. Receiving maximally-tolerated medical therapy for heart failure as indicated per ACC/AHA or ESC Heart Failure Guidelines (guideline-directed medical therapy or GDMT), in the absence of contraindications and lack of availability. GDMT refers to those guideline-directed medical therapies having a Class I indication for use.

   * For patient with heart failure and a reduced ejection fraction (HFrEF), GDMT includes a diuretic as needed for volume control, angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB) or angiotensin receptor neprilysin inhibitor (ARNI), beta-blocker (BB), mineralocorticoid receptor antagonist (MRA), and SGLT2 inhibitor for at least 3 months prior to the Baseline visit. Drug doses, with the exception of diuretics, should be stable for at least 1 month, where stability is defined as no more than a 100% increase or 50% decrease in dose.
   * For patient with heart failure and a preserved ejection fraction (HFpEF), GDMT includes a diuretic as needed for volume control and treatment of associated conditions (e.g., hypertension, atrial fibrillation) for at least 3 months prior to the Baseline visit. Drug doses, with the exception of diuretics, should be stable for at least 1 month, where stability is defined as no more than a 100% increase or 50% decrease in dose.
   * Patients should also receive Class I recommended cardiac rhythm management device therapy. Specifically: if indicated by class I guidelines, cardiac resynchronization therapy (CRT), implanted cardioverter-defibrillator (ICD), or a pacemaker should be implanted at least 3 months prior to Baseline Visit. These criteria may be waived if a patient is clinically contraindicated for these therapies or refuses them and must be attested to by the investigator.
   * GDMT may change over time; the most current versions of the ACC/AHA or ESC Heart Failure Guidelines will supersede the above guidelines.
4. Minimum technological knowledge of either the subject or the caregiver, with a smartphone or tablet for use of the self-management application, including physical ability and access to internet.
5. Provide informed consent for study participation and be willing and able to comply with the required tests, treatment instructions and follow-up visits.

6.5.2. Exclusion criteria

Initial Exclusion Criteria (IEC):

1. Age less than 22 (<22) years old.
2. Subjects who are NYHA class IV and ACC/AHA stage D.
3. Subjects with evidence/history of a major cardiovascular or neurovascular event, such as an intra-cardiac thrombus or history of stroke, transient ischemic attack, systemic or pulmonary thromboembolism, deep vein thrombosis (DVT), within the last 6 months of Baseline Visit.
4. Subjects with a resting systolic blood pressure <90 or >180 mmHg at Baseline Visit.
5. Left ventricular end-diastolic diameter (LVEDD) > 8cm.
6. Have an atrial septal defect or patent foramen ovale with more than trace shunting on color Doppler or intravenous bubble study or surgical or interventional correction of congenital heart disease involving atrial septum, including placement of a PFO or ASD closure device, and have a hypermobile septum or a septal aneurysm.
7. Subjects with untreated severe valve lesions, which are indicated for surgical or percutaneous intervention, active valvular vegetations, atrial myxoma, hypertrophic cardiomyopathy with significant resting or provoked subaortic gradient, acute myocarditis, tamponade, or large pericardial effusion, constrictive pericarditis, infiltrative cardiomyopathy (including cardiac sarcoidosis, amyloidosis, and hemochromatosis), or congenital heart disease, as a cause of HF.
8. Uncontrolled tachyarrhythmia or bradycardia (heart rate <45 bpm).
9. Intractable HF with resting symptoms despite maximal medical therapy (ACC/AHA HF Stage D), including subjects receiving continuous or intermittent outpatient IV vasoactive medications (e.g., IV inotropes, IV vasodilators), or subjects treated with a ventricular assist device (VAD).
10. Intolerant to ACE-I, ARB, or ARNI and beta-blocker medical therapy for subjects classified as HFrEF.
11. The presence of an acute coronary syndrome (ACS), percutaneous coronary intervention (PCI), rhythm management system revision, lead extraction, or cardiac or other major surgery within the preceding 90 days of implant procedure.
12. Subjects not eligible for emergency open-heart, thoracic or vascular surgery.
13. Women who are pregnant or planning to become pregnant.
14. Subjects with a life expectancy that is shorter than 12 months, or those who have received a cardiac transplant or are listed for cardiac transplantation and likely to be transplanted within 12 months of Baseline Visit.
15. Have coagulopathy or uninterruptible anticoagulation therapy or contraindication for all the forms of antiplatelet/anticoagulant treatments anticipated in the protocol.
16. Known history of life-threatening allergy to contrast dye that cannot be properly pre-medicated.
17. Have an estimated Glomerular Filtration Rate (GFR) <25 ml/min/1.73 m2 by the MDRD method or on chronic renal dialysis.
18. Hepatic impairment with at least one liver Function Test (transaminases, total bilirubin, or alkaline phosphatase) ≥ 3 times upper limit of normal.
19. Gastrointestinal bleeding in the last 6 months of implant procedure.
20. Have severe chronic pulmonary disease requiring continuous home oxygen, chronic oral steroid therapy, hospitalization for exacerbation during prior 6 months, or has severe obstructive physiology on PFTs (FEV1/FVC <0.70 and FEV1 < 50% normal), if done.
21. Subjects who have an active infection requiring systemic antibiotics or an elevated white blood count (above the local laboratory reference ranges).
22. Have a history of active drug addiction, active alcohol abuse, or psychiatric hospital admission for psychosis within the prior 2 years.
23. Are currently participating in a clinical study or investigation.
24. Subject otherwise not appropriate for study as determined by the investigator and subjects who are unwilling to comply with the study protocol, or subjects with a history of non-compliance. The reasons must be documented.
25. Subjects contraindicated for trans-septal puncture, TEE or ICE.

    Intra Procedural Exclusion Criteria:

    (Intra Procedural Exclusion Criteria will be determined immediately after intracardiac echocardiography or transesophageal echocardiography determination of left atrial anatomy and just before transseptal puncture)
26. Anatomical anomaly on TEE or ICE that precludes implantation of the V-LAPIM across the interatrial septum (Fossa Ovalis) including: Septal thickness at fossa > 5 mm, FO Dimension <16mm, ASD or PFO with more than a trace amount of shunting, intra-cardiac thrombus felt to be acute and not present on prior exams and abnormal septum, e.g., a hypermobile septum or a septal aneurysm.
27. Inadequate vascular access for implantation of V-LAPIM or are unable to tolerate a right heart catheterization (RHC).
28. Severe pulmonary hypertension at index procedure above 70 mmHg or PVR at index procedure above 4.0 Woods Units (mmHg L-1 min-1), while these cannot be lowered with vasodilators.
29. Resting systolic Blood Pressure <90 or >180 mmHg, not corrected with IV fluid administration or vasodilators.

Ages: 22 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
LAP measurement | Up to 12 months post-procedure
  Freedom from failure of the V-LAP system to obtain LAP measurement from the sensor implant and transmit the LAP data to the V-LAPHCP HCP Interface and the V-LAPPSM Patient Guidance Application up to 12 months post-procedure.
Safety Endpoint - Major Adverse Cardiac and Neurological Events (MACNE) | Up to six months post-procedure
  Number of participants with study (Device and/ or system) related to Major Adverse Cardiac and Neurological Events (MACNE) - as defined in the protocol, as by the independent Clinical Events Committee

SECONDARY OUTCOMES:
Health Care Provider Usability Questionnaire | Up to 24 months post-procedure
  Usability assessment of the V-LAP system will be measured by questionnaires that will be completed by the investigator. Performance Score 1-5 (1=Poor, 5=Excellent)
Target LAP range | Up to 24 months post-procedure
  Ratio (percentage) of follow-up time in the target Left Atrial pressure (LAP) range as defined by the physician.
New York Heart Association (NYHA) functional class | Up to 24 months post-procedure
  Change in NYHA functional class ranking at 6, 12, and 24 months vs. baseline. Stages of Heart Failure scoring 1-4 (1=High, 4=Low)
Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall score | Up to 24 months post-procedure
  Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall score at 6, 12, and 24 months vs. baseline.
  Scores 1-7 (1=Minimum, 7=Maximum)
Patient Global Assessment (PGA) Overall | Up to 24 months post-procedure
  Change in Patient Global Assessment (PGA) Overall score at 6, 12, and 24 months vs. baseline.
  Performance Score -3 - +3 (-3=Poor, +3=Excellent)
Heart failure hospitalization rate | Up to 12months post-procedure
  Heart failure hospitalization rate at 6 and 12 months (rate is calculated as the number of hospitalizations over individual patient follow-up duration).
Heart failure hospitalization duration | Up to 12months post-procedure
  Heart failure hospitalization duration at 6 and 12 months (duration is calculated as number of days hospitalized over individual patient follow-up duration).
Usability Assessment - Patient Usability Questionnaire | Up to 24 months post-procedure
  Usability assessment of the V-LAP system will be measured by questionnaires that will be completed by the patients. Performance Score 1-5 (1=Poor, 5=Excellent)

CONTACTS AND LOCATIONS:
Overall Officials: Rami Kahwash, Prof., Principal Investigator — Ohio State University; Ramesh Emani, Dr., Principal Investigator — Christ Hospital - Linder Research Institute; Sandip Zalawadiya, Dr., Principal Investigator — Vanderbilt University Medical Center; Nir Ayalon, Dr., Principal Investigator — Boston Medical Center; Michael DiVita, Dr., Principal Investigator — NYU Langone
Locations (1):
- One Boston Medical Center Place, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No